CLINICAL TRIAL: NCT05859295
Title: Evaluation of Low-Level Light Therapy on Meibomian Glands Study
Acronym: ELOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: University of Louisville (Other)
Responsible Party: Principal Investigator, Eric R. Ritchey, Assistant Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00004024
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye
Keywords: Meibomian glands; meibomian gland dysfunction; tears
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes; Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low-Level Light Therapy (Other): All subjects will receive 3 15-minute treatments of low level light therapy
  Interventions: Device: Red Low-Level Light Therapy

INTERVENTIONS:
Device: Red Low-Level Light Therapy — Visible red light (633nm) projected onto the face using an light emitting diode (LED) mask
  Other Names: Marco Equinox

SUMMARY:
The goal of this clinical trial is to examine the effect of low-level light therapy (LLLT) on meibomian gland dysfunction and dry eye disease. The main questions it aims to answer are:

1. Does low-level light therapy reduce levels of pro-inflammatory proteins in meibum
2. Does low-level light therapy increase the ratio of non-polar lipids to polar lipids in meibum

Participants will receive 3 15-minute sessions of low-level light therapy. Meibum will be collected before the first treatment and after the final treatment.

DETAILED DESCRIPTION:
Low-level light therapy (LLLT) is a treatment for meibomian gland dysfunction. The proposed mechanism of action is photobiomodulation of cells leading to improved adenosine triphosphate synthesis, reduction of reactive oxygen species in oxidatively-stressed cells, and the activation of transcription factors involved in cellular proliferation, migration and survival. Understanding of how low-level light therapy based therapy alters meibomian gland function is poor. This study will examine the effect of low-level light therapy on individuals with meibomian gland dysfunction. Eligible subjects will receive 15 minutes of low-level light therapy per week over a 3 week period. Meibum collected prior to treatment will be compared to meibum collected after 3 treatment sessions for alteration in protein and lipid composition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at enrollment
* Individuals with mild to moderate meibomian gland dysfunction based on clinical signs, e.g., meibum quality score of 1-3, meibography score of 1, 2, or 3 on the Pult Meiboscale, non-invasive 1st tear break up time of 10 seconds or less, or an Ocular Surface Disease Index (OSDI) score of 13 to 32 points

Exclusion Criteria:

* History of systemic disease associated with aqueous-deficient dry eye disease (e.g., Sjogren's syndrome)
* History of corneal surgery, refractive surgery, eyelid surgery or ocular trauma within 6 months
* History of LipiFlow, iLux, Meiboflow, Intense Pulsed Light (IPL) or low level light therapy (LLLT) within the last 12 months
* Use of photosensitizing medications
* Pregnant and/or lactating females
* Pigmented lesions, tattoos, or skin cancer in the periocular region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Meibum protein composition | 3 weeks
  Proteomic analysis of meibum collected before and after low level light therapy

SECONDARY OUTCOMES:
Meibum lipid composition | 3 weeks
  Lipidomic analysis of meibum collected before and after low level light therapy

OTHER OUTCOMES:
Non-invasive tear break up time | 3 weeks
  Videokeratoscope assessment of time to break up of the tear film
Tear lipid layer thickness | 3 weeks
  Interferometric assessment of the tear film lipid layer
Tear meniscus height | 3 weeks
  Videokeratoscope assessment of the tear meniscus

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Ritchey, OD, PhD, Principal Investigator — The University of Houston College of Optometry
Locations (1):
- The University of Houston College of Optometry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No